CLINICAL TRIAL: NCT05564988
Title: Chronic Remote Ischemic Preconditioning as a Complement to Conventional Prenatal Care for Preeclampsia: a One-center Prospective Randomized Study for Women With Non-severe Preeclampsia Between 24 and 37 Weeks' Gestation
Brief Title: Chronic Remote Ischemic Preconditioning as a Complement to Conventional Prenatal Care for Preeclampsia
Acronym: RIPC
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: DAVID DESSEAUVE (Other)
Responsible Party: Sponsor-Investigator, DAVID DESSEAUVE, Head of delivery room, Centre Hospitalier Universitaire Vaudois
Organization: Centre Hospitalier Universitaire Vaudois (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2021-01516
Record Dates: First submitted 2022-09-26; First posted 2022-10-04 (Actual); Last update posted 2022-10-04 (Actual); Status verified 2022-09

CONDITIONS: Preeclampsia
Keywords: Preconditioning
MeSH Terms: conditions — Pre-Eclampsia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Preconditionning (Experimental): Ischemia will be obtained after inflating the cuff to a pressure of 200 mmHg (or a pressure at least 50 mmHg above the patient's systolic pressure). After a five-minute period, the cuff will be deflated and the arm allowed to reperfuse for five minutes. These maneuvers will be repeated until 3 cycles of ischemia- reperfusion have been completed once a day. Patients will experiment with this procedure for at least 5 days.
  Interventions: Other: Preconditionning
- Control (No Intervention): For subjects assigned to the control group, the pneumatic cuff is placed around the upper arm, and inflation of a blood pressure to a lower pressure (50mmHg) which will result in no impairment of antegrade flow.

INTERVENTIONS:
Other: Preconditionning — Remote ischemic conditioning will be induced using a Tourniquet cuff applied to the patient's non-dominant arm. The device used will be an Ulrich Kariba machine. A strip of absorbent cotton will be applied to the arm and the tension cuff will be placed over it in a standard way. The systolic pressure and the application time will be set manually.
  Ischemia will be obtained after inflating the cuff to a pressure of 200 mmHg (or a pressure at least 50 mmHg above the patient's systolic pressure). After a five-minute period, the cuff will be deflated and the arm allowed to reperfuse for five minutes. These maneuvers will be repeated until 3 cycles of ischemia- reperfusion have been completed once a day. Patients will experiment with this procedure for at least 5 days.
  Arms: Preconditionning

SUMMARY:
Pre-eclampsia is a disease specific to pregnancy that affects 3-5% of women. It is defined by the appearance of high blood pressure after 20 weeks of amenorrhea associated with the presence of proteins in the urine, dysfunction of organs such as the liver, kidneys, lungs or brain, or dysfunction of the placenta. The cause of this disease is still unclear but it would most likely be a placental origin. Pre-eclampsia is a progressive disease that can lead to important complications. To date, there is no treatment for pre-eclampsia other than childbirth and more particularly placental delivery. Nevertheless, it is possible in some cases to stabilize arterial hypertension and thus to hope for a prolongation of the pregnancy.

Our research project aims to study the effect of preconditioning on blood pressure.

Preconditioning consists of using a blood pressure cuff and inflating it on the upper limb -like during a standard blood pressure measurement- for several minutes followed by a rest period in order to create "ischemia-reperfusion" periods. This technique would allow the release of beneficial substances into the bloodstream that would lower blood pressure. This method has been used for several years in different specialties and has produced good results on the heart, kidneys, lungs and brain.

With this technique we hope to stabilize or even reduce blood pressure in cases of pre-eclampsia and thus prolong the pregnancy.

ELIGIBILITY:
Inclusion Criteria:

* Singleton pregnancy
* Gestational age between 24 0/7 and 36 6/7 weeks' gestation
* Hospitalization for non-severe pre-eclampsia (non-severe hypertension = Systolic blood pressure between 140 and 160mmHg, diastolic blood pressure between 90 and 110mmHg associated with one of these: proteinuria >=300mg/24h/thrombocytopenia 100-150G/L/central symptoms such as headache responding to standard analgesics/hyperreflexia without clonus/decreased fibrinogen/haptoglobin <0.1/utero-placental dysfunction with IUGR and/or umbilical Doppler Class II)
* Maternal age >18 years
* Good comprehension of French allowing easy understanding of the information protocol and the consent form

Exclusion Criteria:

* Chronic hypertension
* Renal disease
* Pre-pregnancy diabetes
* Autoimmune disease (SAPL, SLE, Sjögren)
* Severe PE (Systolic blood pressure >160mmHg, diastolic blood pressure >140mmHg, hepatic cytolysis at twice the norm, right hypochondrium or epigastric pain, central symptoms such as clonus or headache resistant to usual treatment or disturbed consciousness, thrombocytopenia <100G/L, acute pulmonary edema, renal failure defined by doubling of baseline creatinine value or creatinine >97 micromol/L)
* Suspected fetal anomaly or malformation
* HELLP syndrome
* Eclampsia attack
* Pathological fetal monitoring
* Known maternal upper limb vascular anomaly
* Severe maternal cardiac pathology
* Maternal history of deep vein thrombosis of the upper limb

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Estimated)
Dates: Start 2022-10 (Estimated); Primary Completion 2025-10 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Decrease blood pressure | Up to 13 weeks
  Comparison of mean of decrease in systolic and diastolic blood pressure (intervention vs placebo) between day 1 and day 5 using ANOVA test
Decreased blood pressure patients | Up to 13 weeks
  Comparison of the number of patients who significantly decreased blood pressures (≥6%), Chi-squared test or Fisher exact test if appropriate

SECONDARY OUTCOMES:
SFLT/PLGF change | Up to 13 weeks
  Comparison of mean change in the SFLT/PLGF ratio
Uterine artery resistance index change | Up to 13 weeks
  Comparison of mean change in the uterine artery resistance index (using ANOVA test)

CONTACTS AND LOCATIONS:
Overall Officials: Hélène Legardeur, Principal Investigator — CHUV

IPD SHARING:
Plan to Share IPD: No